CLINICAL TRIAL: NCT04845373
Title: The Effect of Mediterranean Diet and Low Fat Diet on Hepatic Fat, Inflammation and Oxidative Stress in Obese Adolescents With Nonalcoholic Fatty Liver Disease
Brief Title: Effect of Mediterranean Diet in Obese Adolescents With Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, GAMZE YURTDAŞ, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 47/2020-05
Record Dates: First submitted 2020-11-13; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterrenean diet (Experimental): Mediterranean diet:Target macronutrient energy contributions were 40% from carbohydrate, 35%-40% from fat (with <10% of energy as saturated fat), and 20% of energy as protein.Participant in this group were trained to consume fish, legumes at least 2-3 times a week, walnuts and olive oil every day in accordance with the Mediterranean diet model.
  Interventions: Other: Mediterranean diet
- Low fat diet (Active Comparator): Low fat diet:Target macronutrient energy contributions for the low fat diet diet were 50-60% from carbohydrate, <30% from fat (with <10% of energy as saturated fat), and 20% from protein.Participants in this group were especially recommended to consume low-fat foods.
  Interventions: Other: Control diet: Low fat diet

INTERVENTIONS:
Other: Mediterranean diet — Diet intervention:Mediterranean diet
  Arms: Mediterrenean diet
Other: Control diet: Low fat diet — Low fat diet
  Arms: Low fat diet

SUMMARY:
The aim of this study was to evaluate the effects of mediterranean and low-fat diet on hepatic fat, inflammation markers and oxidative stress in adolescents with nonalcoholic fatty liver disease. This randomized, single-blind controlled study conducted with obese adolescents aged 11-18 years who were admitted to Tepecik Training and Research Hospital Pediatric Gastroenterology Outpatient Clinic with the diagnosis of nonalcoholic fatty liver disease. Participants were randomly assigned to the Mediterranean diet or low-fat diet group.

DETAILED DESCRIPTION:
This study was conducted to evaluate the effect of Mediterranean and low-fat diet on hepatic fat, inflammation and oxidative stress in obese adolescents with nonalcoholic fatty liver disease (NAFLD). The study, which was designed as a single blind randomized control, was completed with 44 obese adolescents diagnosed with NAFLD between the ages of 11-18. Adolescents were randomized to either a Mediterranean diet (n = 22) or a low-fat diet (control diet) (n = 22) for 12 weeks. At the beginning of the study and at the 12th week, adolescents' blood samples, physical activity and food consumption records were taken, anthropometric measurements and body composition analyzes were made, and antioxidant food consumption frequency and Mediterranean diet quality index questionnaire were applied to adolescents. In the controls performed at the 2th, 4th, 6th, 8th, and 10th weeks, the physical activity and food consumption records of the adolescents were repeated and anthropometric measurements and body composition analyzes were made again.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 11-18
* Being obese (BMI ≥95.persentil)
* Getting a diagnosis of Grade≥1 NAFLD

Exclusion Criteria:

* Existence of liver disease (wilson,hepatitis etc.) other than NAFLD
* Drinking alcohol
* Having a history of type 1 and type 2 diabetes
* Using drugs that can cause steatosis
* Using lipid-lowering drugs
* Using weight loss medications
* Having applied dietary therapy for any disease and weight loss
* Existence of a chronic inflammatory disease
* Existence of cancer
* Thyroid dysfunction (hyperthyroid and hypothyroidism)
* Existence of a history of hepatic virus infection
* Having a history of parenteral nutrition
* Being pregnant and breastfeeding
* Receiving antibiotic treatment within 3 months prior to the study
* Regularly consuming foods containing probiotic and prebiotic properties and / or using nutritional supplements

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
Changes in hepatic steatosis | Baseline and week 12
  Hepatic steatosis was evaluated according to liver ultrasonography records during the routine controls of all patients.
Changes in Inflammatory Parameters | Baseline and week 12
  Measurement of serum cytokines levels (C-reaktive protein (CRP), IL-10, IL-6, IL-8, IL-1 beta, TNF-alpha
Changes in oxidative stress markers | Baseline and week 12
  Measurement of oxidative stress markers (Total Antioxidant Status (TAS), Total Oxidant Status (TOS), Paraoxonase Enzyme Activity (PON-1), Total Thiol, Native Thiol, Superoxide Dismutase (SOD), oxidized-LDL, Glutathione peroxidase,Malondialdehyde (MDA), Glutathione (GSH), non-esterified fatty acids (NEFA))
Changes in glycemic profile | Baseline and week 12
  Measurement of fasting glucose, insulin, HbA1c and calculation of HOMA-IR
Changes in liver function tests | Baseline and week 12
  Measurement of Alanine transaminase (ALT),Aspartate transaminase (AST),Gamma-glutamyltransferase (GGT),Alkaline phosphatase (ALP)

SECONDARY OUTCOMES:
Changes in serum cholesterol levels | Baseline and week 12
  Measurement of total cholesterol, LDL, HDL cholesterol
Changes in triglycerides | Baseline and week 12
  Measurement of serum triglyceride (mg/dl)
Changes in blood pressure | Baseline and week 12
  Measurement of systolic and diastolic blood pressure (mm Hg)
Changes in waist, hip and neck circumference | baseline, week 2, week 4, week 6, week 8, week 10 and week 12
  Measurement of waist circumference (cm)
Changes in Body Fat | baseline, week 2, week 4, week 6, week 8, week 10 and week 12
  Measurement of % body fat with BIA
Changes in BMI | baseline, week 2, week 4, week 6, week 8, week 10 and week 12
  weight and height will be measured to report BMI in kg/m2
Changes in some adipokines | Baseline and week 12
  Measurement of serum leptin and adiponectin

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yurtdas G, Akbulut G, Baran M, Yilmaz C. The effects of Mediterranean diet on hepatic steatosis, oxidative stress, and inflammation in adolescents with non-alcoholic fatty liver disease: A randomized controlled trial. Pediatr Obes. 2022 Apr;17(4):e12872. doi: 10.1111/ijpo.12872. Epub 2021 Dec 8. PMID 34881510